CLINICAL TRIAL: NCT00543764
Title: Intraoperative Pathway in DIEP Flap Breast Reconstruction
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Bernard T. Lee, Assistant Professor in Surgery, Beth Israel Deaconess Medical Center
Other Study IDs: 2007-P-000266/1
Record Dates: First submitted 2007-10-12; First posted 2007-10-15 (Estimated); Results first posted 2012-07-06 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-02

CONDITIONS: Breast Cancer
Keywords: Intraoperative Pathway; Breast Reconstruction; DIEP flap
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pre pathway: Pre pathway
- Post pathway: Post pathway
  Interventions: Other: pathway

INTERVENTIONS:
Other: pathway — Comparison of pre and post pathway
  Other Names: intraoperative pathway
  Groups: Post pathway

SUMMARY:
Efficiency in the operating room can be difficult in long cases with multiple surgeons. We used a team based approach to develop an intraoperative pathway for microsurgical breast reconstruction with a deep inferior epigastric perforator flap.

DETAILED DESCRIPTION:
A team based approach was developed with an intraoperative pathway for microsurgical breast reconstruction with a deep inferior epigastric perforator flap.

ELIGIBILITY:
Inclusion Criteria:

* All cases prior to pathway

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing breast reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2005-01; Primary Completion 2008-12 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard T Lee, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2006-2008. Operating room records
Groups:
- Pre Pathway: Patients prior to pathway implementation
- Post Pathway: Patients after pathway implementation
Period: Overall Study
Arm/Group | Pre Pathway | Post Pathway
Started | 100 | 50
Completed | 100 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre Pathway | Post Pathway | Total
Number analyzed (Participants) | 100 | 50 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 100 | 50 | 150
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: paticipants]
  Female | 100 | 50 | 150
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Operative Time
Description: Length of Time in surgery
Time Frame: 3 years
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Pre Pathway | Post Pathway
Number analyzed (Participants) | 100 | 50
hours | 8.2 [7.8 to 8.6] | 6.9 [6.3 to 7.5]

ADVERSE EVENTS:
Arm/Group | Pre Pathway | Post Pathway
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/50
Other Adverse Events (participants affected / at risk) | 0/100 | 0/50

LIMITATIONS AND CAVEATS:
More patient enrollment is necessary to ascertain long term outcomes

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No